CLINICAL TRIAL: NCT05807867
Title: RCT of an Intersectional Stigma Intervention to Sustain Viral Suppression Among Women Living With Serious Mental Illness and HIV in Botswana
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: University of Pennsylvania (Other); University of Botswana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R01TW012402 (NIH)
Record Dates: First submitted 2022-11-23; First posted 2023-04-11 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-07

CONDITIONS: Hiv; Serious Mental Illness
Keywords: HIV; Stigma
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Intervention Model Description: 1. Recruit 180 women to allow for 8% attrition post-intervention, with an added 8% during 4-month follow-up (below), to yield a final sample of N=151 expected to complete WMM or control (n=75 in each of 2 arms).
  2. The investigators expect to recruit ~180 family members to allow for 16% attrition overall, to yield a final sample of N=151 expected to complete the stigma intervention or control (n=75 in each of the 2 arms, under assumption that attrition on average occurs at the same rate in each arm).
Who Masked: Outcomes Assessor
Masking Description: Staff assessing all outcomes will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WMM-based intersectional stigma intervention (Experimental): N=90 Women with SMI and HIV in arm 1 will receive WMM stigma intervention as clients transition from psychiatric hospitalization to outpatient care. The curriculum, co-led by a trained clinician and a peer woman with SMI and HIV, will comprise of 8 group sessions at ~60 minutes each. Following psychiatric stabilization, but while still an inpatient, women participants will receive 5 (delivered 2x weekly) of 8 session anti-stigma intervention. To facilitate community integration, the final 3 WMM-based intervention sessions will be delivered once every two weeks at a community-based setting in Gabarone.
  Parallel Group Stigma intervention: N=90 Family members will receive an adapted 3-session WMM-based group intervention that uses the same intervention components. The first 2 sessions will be held weekly in a private room at Sbrana Hospital, while the final session will be held 2 weeks following client discharge in the same community-based setting as above.
  Interventions: Behavioral: WMM-based intersectional stigma intervention
- Attention placebo control (Active Comparator): To isolate intervention effects, our attention control is designed to mimic all salient features of the WMM-based intervention (i.e., group format, co-leaders, duration, inpatient followed by community location) except for the WMM stigma content. Control co-leaders will receive a 1-day training on the control manual and facilitation techniques. Sessions will focus on general health education (i.e., diet, exercise, avoiding alcohol, and healthy sleep habits) for women with SMI and HIV adapted from Ministry of Health materials. The investigators will offer in-person sessions including facilitated discussions to encourage interaction (per the WMM intervention). The investigators expect participation in the attention control arm (~84% retention) to approximate that of women (and family members) attending the intervention arm. While intended to be salient to women participants and their family members, this program should not decrease stigma nor has it been shown to impact MH outcomes.
  Interventions: Behavioral: Attention placebo control

INTERVENTIONS:
Behavioral: WMM-based intersectional stigma intervention — Intervention components consist of:
  1. psychoeducation: facilitating the achievement of "good womanhood" by adhering to psychiatric medications and ART post-discharge
  2. cognitive restructuring to challenge stereotypes: involves reframing psychiatric and ART adherence postdischarge as enacting 'good womanhood' by countering stereotypes of being unable to care for the family or be a suitable marriage partner
  3. Coping skills for discrimination: promoting safe disclosure of SMI and/or HIV status to facilitate psychiatric and ART adherence post-discharge.
  Note: "enhancing skills for discrimination" sessions for women and family members are provided when female participants transition to outpatient care, thus enabling practice of skills in community-based situations. Intervention closes with a ceremony intended to convey WMM by bestowal of ceremonial shawls. The family member version will follow the same format, but each component will be covered in one session (3 sessions total).
  Arms: WMM-based intersectional stigma intervention
Behavioral: Attention placebo control — To isolate intervention effects, our attention control is designed to mimic all salient features of the WMM-based intervention (i.e., group format, co-leaders, duration, inpatient followed by community location) except for the WMM stigma content.
  Arms: Attention placebo control

SUMMARY:
The study goal is to promote viral load suppression among women with serious mental illness (SMI) and HIV in Botswana, given that these women are especially vulnerable to psychiatric medication nonadherence and symptom exacerbation, which are made worse by stigma and threaten antiretroviral therapy (ART) adherence.

The investigators propose to test an intervention to reduce stigma due to the statuses of SMI and HIV, against an attention control condition, in the high-risk transition period after discharge from an initial psychiatric hospitalization. Specifically, the investigators are conducting a two-arm randomized controlled trial (RCT) with a 4-month follow-up to compare the effectiveness of 1) What Matters Most (WMM)-based intersectional stigma intervention delivered as clients transition from psychiatric hospitalization to outpatient care; and 2) an attention placebo control condition that follows a similar format to isolate the effects of the intervention.

The investigators will also assess policymaker workshops where peer women with SMI and HIV co-lead the reporting of RCT findings via lived experience to policymakers to initiate structural change.

Enabling women with SMI and HIV to resist stigma has the potential to improve their HIV outcomes and empower these women to elicit broader, structural-level change.

DETAILED DESCRIPTION:
The proposed project, "RCT of an intersectional stigma intervention to sustain viral suppression among women living with serious mental illness and HIV in Botswana," will test a culturally tailored stigma intervention among women with co-occurring serious mental illness (SMI) and HIV receiving inpatient treatment at Sbrana Psychiatric Hospital in Lobatse, Botswana, who are then discharged into outpatient care. The culturally tailored stigma intervention is based on our novel 'what matters most' (WMM) approach to target intersectional stigma. The investigators will also be conducting a family-level stigma intervention to test its efficacy at reducing family-level SMI and HIV stigma, and to test family-level stigma as a mechanism for change in VL among women. Lastly, the investigators will pilot a policymaker workshop intended to facilitate structural-level change.

Populations included in the study:

1. Women with SMI and HIV,
2. Family members, and
3. Policymakers and other stakeholders

RESEARCH AIM 2.

The investigators propose a two-arm randomized controlled trial (RCT) with a 4-month follow-up to compare the effectiveness of our WMM-based stigma intervention to reduce viral load (VL) at 4-month follow-up (primary outcome) and improve the secondary outcomes of antiretroviral treatment (ART) and psychiatric treatment adherence, MH outcomes (e.g., depression), and social outcomes (e.g., social integration).

In Botswana, families are usually contacted and engaged in psychiatric treatment planning during inpatient stay or on admission. The involvement of family continues during outpatient follow-ups since most patients are accompanied by some relative or caregiver on such visits. Because family acceptance can bolster achieving the capabilities of 'good womanhood' (i.e., by being a family caregiver), family members will receive a parallel, group stigma intervention, which could further facilitate treatment adherence of the recently discharged family member. Therefore, the investigators will conduct a parallel two-arm intervention among women's family members to test its effectiveness in reducing family-level stigma and to assess family-level stigma as a mechanism of change for primary and secondary outcomes among women with SMI and HIV (e.g., VL, ART and psychiatric treatment adherence, MH outcomes and Social outcomes).

Participants in Research Aim 2 will be 75% female identified (100% of inpatient participants will be female-identified, and the investigators are accounting for a 50-50 gender split among recruited family members). Estimated distribution is 270 women, 90 men.

* Recruit 180 women to allow for 8% attrition post-intervention, with an added 8% during 4-month follow-up (below), to yield a final sample of N=151 expected to complete WMM or control (n=75 in each of 2 arms).
* The investigators expect to recruit ~180 family members to allow for 16% attrition overall, to yield a final sample of N=151 expected to complete the stigma intervention or control (n=75 in each of the 2 arms, under assumption that attrition on average occurs at the same rate in each arm).

RESEARCH AIM 3.

The investigators further propose to pilot and evaluate policymaker workshops whereby peer women with SMI and HIV share RCT findings via lived experience to policymakers to initiate structural-level change.

The investigators anticipate that the multisectoral stakeholder committee members (n=15) and policymakers (n=50) in Research Aim 3 will have ~50-50 gender split - 32 women, 33 men.

* The investigators plan to convene a Multisectoral Stakeholder Committee facilitate development of the policymaker workshops. Our MSC will include policymakers across multiple sectors: Ministry of Health (MoH), District Health Management Team (DHMT), Policy, Academic leaders
* The investigators additionally plan to recruit 50 policy makers to participate in the policymaker workshops in conjunction with 2-3 peer co-leader women with SMI and HIV to reduce stigma among policymakers and lay a foundation for sustaining interventions to improve HIV and other health outcomes in this vulnerable group.

OVERVIEW.

UBotswana will recruit participants and conduct the intervention, assessments, and data management. Overseen by PI Yang, NYU will provide study oversight, expertise in WMM and stigma, and conduct data analyses; UPenn will provide expertise in integration of the intervention for SMI and HIV; Botswana-UPenn Partnership will provide expertise in integration of peers into stigma interventions and implementation of community based interventions in Botswana; UCSF and UC Riverside will offer expertise and supervision in stigma interventions.

ELIGIBILITY:
(A) WOMEN WITH SMI AND HIV

At Sbrana Psychiatric Hospital, the investigators will recruit women with SMI and HIV who are receiving treatment at that facility. Women with SMI and HIV will be receiving psychiatric care and ART and must:

1. Meet DSM-5 criteria for current psychotic disorder or mood disorders or other disorders causing functional impairment except substance use disorders and developmental disorders, per clinician interview based on the MINI
2. Have confirmed HIV positive status
3. Be 18-55 years of age
4. Be female
5. Have capacity to provide consent and written informed consent
6. Speak English or Setswana
7. Be a Botswana citizen

   The investigators will also recruit 6 to 8 women with SMI and HIV as peer co-leaders to facilitate the intervention. For women who are peer co-leaders, inclusion criteria include #1 to #7 above in addition to:
8. Remaining adherent to psychiatric medications
9. Being symptomatically stable for >2 years
10. Maintaining consistent ART adherence.

(B) FAMILY MEMBERS OF WOMEN WITH SMI AND HIV.

In Botswana, families are usually contacted and engaged in psychiatric treatment planning during inpatient stay or on admission. The involvement of family continues during outpatient follow-ups since most patients are accompanied by some relative or caregiver on such visits. Eligible participants include:

1. Identified by participant and/or clinician as the relative 'most involved in the client's care'.
2. Be 18-65 years of age
3. English or Setswana speaking
4. Botswana citizen.

(C) POLICY MAKERS AND OTHER STAKEHOLDERS.

Policy makers will be

1. Be 18-55 years of age
2. Include: (a) bureaucratic officials of Botswana, public sector ministries (government) at the national level holding appointment to senior offices that develop, interpret and/or implement national mental health and HIV programs (prevention and treatment) or related clinical services; (b) senior bureaucratic officials of the National AIDS and Health Promotion Agency (NAHPA); and (c) senior members of civil society organizations (CSOs), nongovernment organizations (NGOs) or other entities that support the national Botswana government to implement services to People Living With HIV (PLWH) and mental health patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Viral load (VL) | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  1) Blood draw: VL deﬁned dichotomously (0=<25 copies/mL, 1= >25 copies/mL) and continuously (log transformed)
Viral load | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  2) Medical records: Routine & month VL monitoring at IDCC

SECONDARY OUTCOMES:
Mental Health (MH) and Social outcomes | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) PRIME screen: psychosis,12 items
Mental Health (MH) and Social outcomes | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) CES-D: depressive symptoms, 20 items
Mental Health (MH) and Social outcomes | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) GAD-7: Anxiety symptoms, 7 items
Mental Health (MH) and Social outcomes | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) PCL-5: trauma symptoms, 20 items
Mental Health (MH) and Social outcomes | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) ISEL: social support, 4x 10 item subscales eg. belonging
Mental Health (MH) and Social outcomes | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) Social integration scale: community integration, 10 items
Mental Health (MH) and Social outcomes | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) EQ5D: health related quality of life, 5 items
Psychiatric adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  1) Self report: Medication Adherence Rating Scale (MARS): attitudes and behaviors reflecting members' psychiatric medication adherence, 10 items
Psychiatric adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  2) Chart review: adherence to psychiatric outpatient appointments
ART adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Medical records) : Refill monitoring via pharmacy records
ART adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) AACTG Adherence Instrument: AACTG Adherence instrument, 3 items
ART adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (EHR) : facility-records of HIV visits

OTHER OUTCOMES:
Women's stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) Kalichman HIV Stigma Scale: Internalized stigma e.g. HIV disclosure; 6 items
Women's stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) Berger HIV Stigma Scale: perceived community stigma, anticipated stigma, enacted stigma; 27 items
Women's stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) Internalized stigma of mental illness scale: 3 subscales (a) discrimination experience 5 items, (b) alienation 6 items, (c) social withdrawal 6 items
Women's stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) Gender-Equitable Scale: attitudes towards gender norms e.g. sexuality; 4 subscales, 24 items
Women's stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) WMM Womanhood + HIV: Culture Shapes, Culture Protects subscales; 20 items
Women's stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) WMM Womanhood + SMI: Scale items to be developed in Aim 1
Family members' stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) Devaluation of families scale: family members' experience of SMI stigma, 7 items
Family members' stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) Courtesy Stigma Scale: family members' experience of HIV stigma; 9 items
Family members' stigma | Changes from baseline at 4 months after intervention completion (approximately 16 months from baseline)
  (Self-report) Gender-Equitable Scale: attitudes towards gender norms e.g. sexuality; 4 subscales, 24 items
Other Covariates for women with SMI and HIV: HIV Treatment adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) distance to clinic; when ART initiated; side effect profile; 3 items
Other Covariates for women with SMI and HIV: Psychiatric Treatment Adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) distance to clinic; visits to spiritual/traditional healers (Y/N and # of visits)
Other Covariates for women with SMI and HIV: Psychiatric Treatment Adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) Beck Cognitive Insight Scale: illness insight; 15 items
Other Covariates for women with SMI and HIV: Psychiatric Treatment Adherence | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) psychiatric medication side effects
Other Covariates for women with SMI and HIV: Gender-based behaviors & experiences | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) HIV Risk-Taking Behavior Scale: sexual risk behaviors; 11 items
Other Covariates for women with SMI and HIV: Gender-based behaviors & experiences | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) Woman Abuse Screening: IPV; 8 items
Other Covariates for women with SMI and HIV: Social desirability | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) Marlowe-Crowne Social Desirability Scale: 13 items
Other Covariates for family members: Subjective family burden inventory scale | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) Zarit Burden Interview: family burden: subjective; 22 items
Other Covariates for family members: Causal model subscales | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) Causal Model Questionnaire for Schizophrenia: 6 subscales assessing explanatory model for SMI
Sociodemographics for women with SMI and HIV | Baseline
  (Self-report) : age; education; employment; income; marital status; urban/rural residence; living with family; maternal status; # of children; religiosity/religious affiliation
Clinical characteristics for women with SMI and HIV | Baseline
  (Self-report) : onset age of psychiatric symptoms; duration of psychiatric illness; first psychiatric tx contact; diagnosis (psychotic/bipolar/severe depression); first diagnosis of HIV; first HIV treatment
Clinical characteristics for women with SMI and HIV- Alcohol use | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) AUDIT: alcohol use, 10 items
Clinical characteristics for women with SMI and HIV- Substance use | Changes from baseline to intervention completion (an average of 12 months), and to 4 months (or 16 months from baseline) after intervention completion
  (Self-report) DUDIT: substance use, used with AUDIT, 11 items
Sociodemographics and clinical characteristics for family members | Baseline
  (Self-report) : Age; gender; education; income/employment; relationship to patient; religiosity/religious affiliation; HIV status; previous psych diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Yang, PhD, Principal Investigator — New York University
Locations (1):
- Princess Marina Hospital IDCC, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.